CLINICAL TRIAL: NCT04510922
Title: Technology-Based Objective Measures for Gait and Postural Assessment in Parkinson Disease Patients With Orthostatic Hypotension: Feasibility and Effect-Size Finding Study
Brief Title: Lundbeck TOMs Orthostatic Hypotension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alberto Espay, MD, MSc (Other)
Collaborators: Lundbeck LLC (Industry)
Responsible Party: Sponsor-Investigator, Alberto Espay, MD, MSc, Professor of Neurology, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Lundbeck-TOMs-OH-001
Record Dates: First submitted 2020-07-09; First posted 2020-08-12 (Actual); Results first posted 2022-09-26 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-08

CONDITIONS: Orthostatic Hypotension; Idiopathic Parkinson Disease
MeSH Terms: conditions — Hypotension, Orthostatic; Parkinson Disease | interventions — Droxidopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Droxidopa (Experimental): 100-600mg droxidopa TID
  Interventions: Drug: Droxidopa 100 MG [Northera]

INTERVENTIONS:
Drug: Droxidopa 100 MG [Northera] — droxidopa taken three times a day titrated up to a maximum of 600 mg.

SUMMARY:
Orthostatic hypotension (OH), which consists in a significant reduction in blood pressure levels upon standing from a seated position, may affect approximately one in three patients with Parkinson's disease (PD). It usually presents as dizziness, lightheadedness, feeling faint, or feeling like you might black out while standing. This can significantly impact the quality of life (QoL) of PD patients, resulting in difficulties with balance, walking, and increased risk of falls. The main aim of this study is to evaluate whether the use of technological devices (a computerized system for analyzing abnormalities in walking in clinical settings and a wearable sensor to detect changes in postural unsteadiness in the home environment) may improve the detection of complications and the response to medical therapies for OH in patients with PD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's Disease, meeting UK Brain Bank criteria for at least 3 years
* Hoehn and Yahr (H&Y) stage I-III
* Age between 30 and 80 years old (both inclusive)
* Stable dosage of dopaminergic medications for at least 4 weeks
* Orthostatic Hypotension, defined as a fall in systolic BP ≥ 20 mmHg or diastolic BP ≥ 10 mmHg within 3 minutes of standing
* Willingness and ability to comply with scheduled visits

Exclusion Criteria:

* Diabetes mellitus or other diseases potentially associated with autonomic dysfunction
* Treatment with antihypertensive drugs or with alpha-adrenergic antagonists
* Cognitive impairment, defined as a score < 24 at the Montreal Cognitive Assessment (MoCA)
* Any atypical signs lowering the diagnostic certainty for PD
* Lack of postural reflex defined as a score > 2 at the MDS-UPDRS item 3.12 (recover at the pull test)
* Severe levodopa induced dyskinesia, defined as an MDS-UPDRS item 4.2 > 2 (functional impact of dyskinesia)

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Velseboer DC, de Haan RJ, Wieling W, Goldstein DS, de Bie RM. Prevalence of orthostatic hypotension in Parkinson's disease: a systematic review and meta-analysis. Parkinsonism Relat Disord. 2011 Dec;17(10):724-9. doi: 10.1016/j.parkreldis.2011.04.016. Epub 2011 May 14. PMID 21571570
- [Background] Palma JA, Gomez-Esteban JC, Norcliffe-Kaufmann L, Martinez J, Tijero B, Berganzo K, Kaufmann H. Orthostatic hypotension in Parkinson disease: how much you fall or how low you go? Mov Disord. 2015 Apr 15;30(5):639-45. doi: 10.1002/mds.26079. Epub 2015 Feb 12. PMID 25678194
- [Background] Senard JM, Rai S, Lapeyre-Mestre M, Brefel C, Rascol O, Rascol A, Montastruc JL. Prevalence of orthostatic hypotension in Parkinson's disease. J Neurol Neurosurg Psychiatry. 1997 Nov;63(5):584-9. doi: 10.1136/jnnp.63.5.584. PMID 9408097
- [Background] Tan LC, Tan AK, Tjia HT. The profile of hospitalised patients with Parkinson's disease. Ann Acad Med Singap. 1998 Nov;27(6):808-12. PMID 10101555
- [Background] Woodford H, Walker R. Emergency hospital admissions in idiopathic Parkinson's disease. Mov Disord. 2005 Sep;20(9):1104-8. doi: 10.1002/mds.20485. PMID 15884038
- [Background] Vossius C, Nilsen OB, Larsen JP. Parkinson's disease and hospital admissions: frequencies, diagnoses and costs. Acta Neurol Scand. 2010 Jan;121(1):38-43. doi: 10.1111/j.1600-0404.2009.01239.x. Epub 2009 Sep 10. PMID 19744137
- [Background] Kaufmann H, Malamut R, Norcliffe-Kaufmann L, Rosa K, Freeman R. The Orthostatic Hypotension Questionnaire (OHQ): validation of a novel symptom assessment scale. Clin Auton Res. 2012 Apr;22(2):79-90. doi: 10.1007/s10286-011-0146-2. Epub 2011 Nov 2. PMID 22045363
- [Background] Merola A, Romagnolo A, Rosso M, Lopez-Castellanos JR, Wissel BD, Larkin S, Bernardini A, Zibetti M, Maule S, Lopiano L, Espay AJ. Orthostatic hypotension in Parkinson's disease: Does it matter if asymptomatic? Parkinsonism Relat Disord. 2016 Dec;33:65-71. doi: 10.1016/j.parkreldis.2016.09.013. Epub 2016 Sep 10. PMID 27641792
- [Background] Hubble RP, Naughton GA, Silburn PA, Cole MH. Wearable sensor use for assessing standing balance and walking stability in people with Parkinson's disease: a systematic review. PLoS One. 2015 Apr 20;10(4):e0123705. doi: 10.1371/journal.pone.0123705. eCollection 2015. PMID 25894561
- [Background] Tinetti ME. Performance-oriented assessment of mobility problems in elderly patients. J Am Geriatr Soc. 1986 Feb;34(2):119-26. doi: 10.1111/j.1532-5415.1986.tb05480.x. No abstract available. PMID 3944402
- [Background] Jenkinson C, Fitzpatrick R, Peto V, Greenhall R, Hyman N. The Parkinson's Disease Questionnaire (PDQ-39): development and validation of a Parkinson's disease summary index score. Age Ageing. 1997 Sep;26(5):353-7. doi: 10.1093/ageing/26.5.353. PMID 9351479
- [Background] Robbins TW, James M, Owen AM, Sahakian BJ, McInnes L, Rabbitt P. Cambridge Neuropsychological Test Automated Battery (CANTAB): a factor analytic study of a large sample of normal elderly volunteers. Dementia. 1994 Sep-Oct;5(5):266-81. doi: 10.1159/000106735. PMID 7951684
- [Background] Karrasch M, Laatu S, Martikainen K, Marttila R. CERAD test performance and cognitive impairment in Parkinson's disease. Acta Neurol Scand. 2013 Dec;128(6):409-13. doi: 10.1111/ane.12138. Epub 2013 May 14. PMID 23668316
- [Background] Espay AJ, Bonato P, Nahab FB, Maetzler W, Dean JM, Klucken J, Eskofier BM, Merola A, Horak F, Lang AE, Reilmann R, Giuffrida J, Nieuwboer A, Horne M, Little MA, Litvan I, Simuni T, Dorsey ER, Burack MA, Kubota K, Kamondi A, Godinho C, Daneault JF, Mitsi G, Krinke L, Hausdorff JM, Bloem BR, Papapetropoulos S; Movement Disorders Society Task Force on Technology. Technology in Parkinson's disease: Challenges and opportunities. Mov Disord. 2016 Sep;31(9):1272-82. doi: 10.1002/mds.26642. Epub 2016 Apr 29. PMID 27125836
- [Background] Gibb WR, Lees AJ. The relevance of the Lewy body to the pathogenesis of idiopathic Parkinson's disease. J Neurol Neurosurg Psychiatry. 1988 Jun;51(6):745-52. doi: 10.1136/jnnp.51.6.745. PMID 2841426
- [Background] Lahrmann H, Cortelli P, Hilz M, Mathias CJ, Struhal W, Tassinari M. EFNS guidelines on the diagnosis and management of orthostatic hypotension. Eur J Neurol. 2006 Sep;13(9):930-6. doi: 10.1111/j.1468-1331.2006.01512.x. PMID 16930356
- [Background] Dineen J, Freeman R. Autonomic Neuropathy. Semin Neurol. 2015 Aug;35(4):458-68. doi: 10.1055/s-0035-1558983. Epub 2015 Oct 6. PMID 26502768
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Jordan J, Biaggioni I. Diagnosis and treatment of supine hypertension in autonomic failure patients with orthostatic hypotension. J Clin Hypertens (Greenwich). 2002 Mar-Apr;4(2):139-45. doi: 10.1111/j.1524-6175.2001.00516.x. PMID 11927799
- [Background] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984
- [Background] O'Sullivan JD, Said CM, Dillon LC, Hoffman M, Hughes AJ. Gait analysis in patients with Parkinson's disease and motor fluctuations: influence of levodopa and comparison with other measures of motor function. Mov Disord. 1998 Nov;13(6):900-6. doi: 10.1002/mds.870130607. PMID 9827613

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only 9 participants completed the study.
Period: Overall Study
Arm/Group | Droxidopa
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Droxidopa
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Orthostatic Hypotension Questionnaire (OHQ) Score
Description: Orthostatic Hypotension Symptom Assessment (OHSA; Range: 0-10) and Orthostatic Hypotension Daily Activities Scale (OHDAS; Range: 0-10) 10 items measured on a Likert-scale with 10 being the worst possible score.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Droxidopa
Number analyzed (Participants) | 9
score on a scale | 4.6 (1.9)

2. Primary Outcome: Tinetti Score
Description: he Tinetti assessment tool is an easily administered task-oriented test that measures an older adult's gait and balance abilities. Scoring: Items are scored either "0-1" or "0-2". "0" indicates the highest level of impairment, whereas a higher score (1 or 2) indicates the individuals independence.
  There were 17 tasks (one task split into two sub-items and scored twice) that the scores were summed for a highest possible score of 28 (10 items scored on a 0-1 scale, and 8 items scored on a 0-2 scale).
  The Tinetti assessment was compared pre- and post- 6 week medication dosing.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Droxidopa
Number analyzed (Participants) | 9
score on a scale | 13.4 (2.07)

3. Primary Outcome: PDQ-39 Score
Description: The Parkinson's Disease Questionnaire (PDQ-39) assesses how often people with Parkinson's experience difficulties across 8 dimensions of daily living including mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort.
  The scale consists of 39 items ranked on a 5-point ordinal scale (Never=0, Occasionally=1, Sometimes=2, Often=3, Always=4).
  Each dimension total score range from 0 (never have difficulty) to 100 (always have difficulty). Lower scores reflect better Quality of Life.
  Dimension score = sum of scores of each item in the dimension divided by the maximum possible score of all the items in the dimension, multiplied by 100.
  Overall score = sum of dimension total scores divided by 8.
  Scores were compared pre- and post- 6 weeks dosing with medication.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Droxidopa
Number analyzed (Participants) | 9
score on a scale | 31 (18.1)

4. Primary Outcome: Gait Analysis - Stride Length
Description: Measured in cm
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Droxidopa
Number analyzed (Participants) | 9
cm | 60.3 (9)

5. Primary Outcome: Gait Analysis - Single Leg Stance Time
Description: Using a gait mat, participants were instructed to walk self-paced along the mat. The sensors in the mat automatically extracted the percentage of time a participant stood on a single leg. The output was compared pre- and post- 6 week dosing with study medication.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Droxidopa
Number analyzed (Participants) | 9
percentage of time | 34.6 (2)

6. Primary Outcome: Gait Analysis - Gait Velocity
Description: Using a gait mat, participants were instructed to walk self-paced on the mat, turn around, and walk back. Their velocity was measured in cm/sec.
  This output was compared pre- and post- 6 week dosing with study medication.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Droxidopa
Number analyzed (Participants) | 9
cm/sec | 112.1 (17.2)

7. Primary Outcome: Postural Analysis - Postural Sway
Description: Using a gait mat, postural sway was measured in cm on the X-axis while participants were asked to stand eyes open and eyes closed for 30 seconds. This output was compared pre- and post- 6 weeks dosing with study medication.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Droxidopa
Number analyzed (Participants) | 9
cm | 35.8 (51.2)

ADVERSE EVENTS:
Time Frame: Adverse Events were monitored for each participant during the 6 weeks they were enrolled.
Arm/Group | Droxidopa
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-31): https://cdn.clinicaltrials.gov/large-docs/22/NCT04510922/Prot_SAP_000.pdf